CLINICAL TRIAL: NCT03579940
Title: Safety, Tolerability, and Pharmacokinetics of Lasmiditan in Healthy Japanese and Caucasian Subjects
Brief Title: A Study of Lasmiditan in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17010; H8H-JE-LAIE (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-25; First posted 2018-07-09 (Actual); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lasmiditan - Japanese (Experimental): Single (50 milligram (mg), 100 mg, 200 mg, 400 mg) and repeated (2 × 200 mg) doses of Lasmiditan administered orally in up to three of three study periods.
  Interventions: Drug: Lasmiditan
- Placebo - Japanese (Placebo Comparator): Single and repeated (2 X placebo) doses of Placebo administered orally in up to one of three study periods.
  Interventions: Drug: Placebo
- Lasmiditan - Caucasian (Experimental): Single (50 mg, 100 mg, 200 mg) dose of Lasmiditan administered orally in up to three of three study periods.
  Interventions: Drug: Lasmiditan
- Placebo - Caucasian (Placebo Comparator): Single dose of Placebo administered orally in up to one of three study periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144
  Arms: Lasmiditan - Caucasian; Lasmiditan - Japanese
Drug: Placebo — Administered orally.
  Arms: Placebo - Caucasian; Placebo - Japanese

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of lasmiditan in healthy Japanese and Caucasian participants. The study will also investigate how much lasmiditan gets into the bloodstream and how long it takes the body to get rid of lasmiditan when given to Japanese and Caucasians. The study will last up to 47 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy Japanese (first generation) or Caucasian males or females, as determined by medical history and physical examination
* Have a body mass index of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds or any components of the formulation of lasmiditan
* Have previously received the investigational product in this study, withdrawn from this study, or received lasmiditan in any other study investigating lasmiditan
* Have an abnormal supine blood pressure at screening.
* Have a history of syncope, presyncope, uncontrolled vertigo, postural dizziness, or a risk of falls, as judged to be clinically significant by the investigator, or have orthostatic decreases in supine blood pressure of >20 millimeters of mercury (mmHg), or have orthostatic decreases in diastolic blood pressure of >10 mmHg at screening.
* Are women who are pregnant, lactating, or have a positive pregnancy test at screening or admission to the clinical research unit (CRU)
* Have donated blood of more than 500 milliliters (mL) within 1 month prior to screening

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with three study periods, each participant received single/repeated oral doses of 50, 100, 200, 400, or 2 X 200 milligram (mg) lasmiditan, placebo, or 2 X placebo, according to their assigned treatment sequence, on Day 1 of each Period. The washout period between dosing in consecutive study periods was approximately 72 hours.
Groups:
- Cohort 1: Sequence 1: Japanese; Cohort 3: Sequence 1: Caucasian: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo Period 2: 100 mg Lasmiditan and Period 3: 200 mg Lasmiditan.
- Cohort 1: Sequence 2: Japanese; Cohort 3: Sequence 2: Caucasian: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 50 mg Lasmiditan Period 2: Placebo and Period 3: 200 mg Lasmiditan.
- Cohort 1: Sequence 3: Japanese; Cohort 3: Sequence 3: Caucasian: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 50 mg Lasmiditan Period 2: 100 mg Lasmiditan and Period 3: Placebo.
- Cohort 2: Sequence 1: Japanese: Participants received single, repeated oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo Period 2: 400 mg Lasmiditan and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 2: Japanese: Participants received single, repeated oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 50 mg Lasmiditan Period 2: Placebo and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 3: Japanese: Participants received single oral doses of Lasmiditan and repeated oral doses of placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 100 mg Lasmiditan Period 2: 400 mg Lasmiditan and Period 3: 2 X Placebo (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 4: Japanese: Participants received single, repeated oral doses of Lasmiditan on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 200 mg Lasmiditan Period 2: 400 mg Lasmiditan and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Cohort 3: Sequence 4: Caucasian: Participants received single oral doses of Lasmiditan on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 50 mg Lasmiditan Period 2: 100 mg Lasmiditan and Period 3: 200 mg Lasmiditan .
Period: Period 1
Arm/Group | Cohort 1: Sequence 1: Japanese | Cohort 1: Sequence 2: Japanese | Cohort 1: Sequence 3: Japanese | Cohort 2: Sequence 1: Japanese | Cohort 2: Sequence 2: Japanese | Cohort 2: Sequence 3: Japanese | Cohort 2: Sequence 4: Japanese | Cohort 3: Sequence 1: Caucasian | Cohort 3: Sequence 2: Caucasian | Cohort 3: Sequence 3: Caucasian | Cohort 3: Sequence 4: Caucasian
Started | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Received at Least 1 Dose of Study Drug | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Sequence 1: Japanese | Cohort 1: Sequence 2: Japanese | Cohort 1: Sequence 3: Japanese | Cohort 2: Sequence 1: Japanese | Cohort 2: Sequence 2: Japanese | Cohort 2: Sequence 3: Japanese | Cohort 2: Sequence 4: Japanese | Cohort 3: Sequence 1: Caucasian | Cohort 3: Sequence 2: Caucasian | Cohort 3: Sequence 3: Caucasian | Cohort 3: Sequence 4: Caucasian
Started | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 2 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1: Sequence 1: Japanese | Cohort 1: Sequence 2: Japanese | Cohort 1: Sequence 3: Japanese | Cohort 2: Sequence 1: Japanese | Cohort 2: Sequence 2: Japanese | Cohort 2: Sequence 3: Japanese | Cohort 2: Sequence 4: Japanese | Cohort 3: Sequence 1: Caucasian | Cohort 3: Sequence 2: Caucasian | Cohort 3: Sequence 3: Caucasian | Cohort 3: Sequence 4: Caucasian
Started | 3 | 2 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 2 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Cohort 2: Sequence 1: Japanese: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo Period 2: 400 mg Lasmiditan and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 2: Japanese: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 50 mg Lasmiditan Period 2: Placebo and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 3: Japanese: Participants received single oral doses of Lasmiditan and placebo on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 100 mg Lasmiditan Period 2: 400 mg Lasmiditan and Period 3: 2 X Placebo (2 single doses administered 2 hours apart).
- Cohort 2: Sequence 4: Japanese: Participants received single oral doses of Lasmiditan on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 200 mg Lasmiditan Period 2: 400 mg Lasmiditan and Period 3: 2 X 200 mg Lasmiditan (2 single doses administered 2 hours apart).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Sequence 1: Japanese | Cohort 1: Sequence 2: Japanese | Cohort 1: Sequence 3: Japanese | Cohort 2: Sequence 1: Japanese | Cohort 2: Sequence 2: Japanese | Cohort 2: Sequence 3: Japanese | Cohort 2: Sequence 4: Japanese | Cohort 3: Sequence 1: Caucasian | Cohort 3: Sequence 2: Caucasian | Cohort 3: Sequence 3: Caucasian | Cohort 3: Sequence 4: Caucasian | Total
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 27
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 13
  Male | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 1 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: The number of participants with 1 or more SAEs considered by the investigator to be related to study drug administration is reported. Summaries of SAEs and other non-serious adverse events (AEs), regardless of causality, are located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 20
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Japanese; Placebo: Caucasian: Participants received single oral dose of placebo on day 1.
- 2 x Placebo: Japanese: Participants received 2 x Placebo (2 single oral doses administered 2 hours apart) on day 1.
- 50 mg Lasmiditan: Japanese; 50 mg Lasmiditan: Caucasian: Participants received single oral dose of 50 mg lasmiditan on day 1.
- 100 mg Lasmiditan: Japanese; 100 mg Lasmiditan: Caucasian: Participants received single oral dose of 100 mg lasmiditan on day 1.
- 200 mg Lasmiditan: Japanese; 200 mg Lasmiditan: Caucasian: Participants received single oral dose of 200 mg lasmiditan on day 1
- 400 mg Lasmiditan: Japanese: Participants received single oral dose of 400 mg lasmiditan on day 1.
- 2 X 200 mg Lasmiditan: Japanese: Participants received 2 X 200 mg lasmiditan (2 single oral doses administered 2 hours apart) on day 1.
Arm/Group | Placebo: Japanese | Placebo: Caucasian | 2 x Placebo: Japanese | 50 mg Lasmiditan: Japanese | 50 mg Lasmiditan: Caucasian | 100 mg Lasmiditan: Japanese | 100 mg Lasmiditan: Caucasian | 200 mg Lasmiditan: Japanese | 200 mg Lasmiditan: Caucasian | 400 mg Lasmiditan: Japanese | 2 X 200 mg Lasmiditan: Japanese
Number analyzed (Participants) | 10 | 8 | 2 | 6 | 8 | 7 | 8 | 8 | 9 | 7 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Lasmiditan in Each Period
Description: PK: AUC(0-∞) of Lasmiditan in Each Period was evaluated.
Time Frame: Period 1 and Period 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose; Period 3: predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 36 and 48 hours postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 50 mg Lasmiditan: Japanese | 50 mg Lasmiditan: Caucasian | 100 mg Lasmiditan: Japanese | 100 mg Lasmiditan: Caucasian | 200 mg Lasmiditan: Japanese | 200 mg Lasmiditan: Caucasian | 400 mg Lasmiditan: Japanese | 2 X 200 mg Lasmiditan: Japanese
Number analyzed (Participants) | 6 | 8 | 7 | 8 | 8 | 9 | 7 | 7
nanogram*hour per milliliter (ng*h/mL) | 362 (46) | 366 (78) | 791 (22) | 826 (70) | 1540 (26) | 2120 (50) | 3780 (32) | 3500 (26)

3. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Lasmiditan in Each Period
Description: PK: Cmax of Lasmiditan in Each Period was evaluated.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 50 mg Lasmiditan: Japanese | 50 mg Lasmiditan: Caucasian | 100 mg Lasmiditan: Japanese | 100 mg Lasmiditan: Caucasian | 200 mg Lasmiditan: Japanese | 200 mg Lasmiditan: Caucasian | 400 mg Lasmiditan: Japanese | 2 X 200 mg Lasmiditan: Japanese
Number analyzed (Participants) | 6 | 8 | 7 | 8 | 8 | 9 | 7 | 7
nanogram per milliliter (ng/mL) | 54.1 (35) | 52.4 (84) | 122 (18) | 101 (94) | 249 (39) | 309 (51) | 680 (40) | 519 (24)

ADVERSE EVENTS:
Time Frame: Up To 20 days
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Placebo: Japanese | Placebo: Caucasian | 2 x Placebo: Japanese | 50 mg Lasmiditan: Japanese | 50 mg Lasmiditan: Caucasian | 100 mg Lasmiditan: Japanese | 100 mg Lasmiditan: Caucasian | 200 mg Lasmiditan: Japanese | 200 mg Lasmiditan: Caucasian | 400 mg Lasmiditan: Japanese | 2 x 200 mg Lasmiditan: Japanese
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/2 | 0/6 | 0/8 | 0/7 | 0/8 | 0/8 | 0/9 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/2 | 0/6 | 0/8 | 0/7 | 0/8 | 0/8 | 0/9 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/10 | 0/8 | 0/2 | 2/6 | 4/8 | 5/7 | 3/8 | 6/8 | 3/9 | 6/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Japanese (N=10) | Placebo: Caucasian (N=8) | 2 x Placebo: Japanese (N=2) | 50 mg Lasmiditan: Japanese (N=6) | 50 mg Lasmiditan: Caucasian (N=8) | 100 mg Lasmiditan: Japanese (N=7) | 100 mg Lasmiditan: Caucasian (N=8) | 200 mg Lasmiditan: Japanese (N=8) | 200 mg Lasmiditan: Caucasian (N=9) | 400 mg Lasmiditan: Japanese (N=7) | 2 x 200 mg Lasmiditan: Japanese (N=7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03579940/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03579940/SAP_001.pdf